CLINICAL TRIAL: NCT06305429
Title: Encouraging Positive Parenting Habits Through Digital Media: Feasibility Study
Brief Title: Encouraging Positive Parenting Habits
Acronym: HABITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Okinawa Institute of Science and Technology Graduate University (Other)
Responsible Party: Principal Investigator, Paulo Eduardo Luiz de Mattos, Researcher, D'Or Institute for Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HABITE
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: ADHD
Keywords: ADHD; Parent Training; Treatment Access
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open, single-group trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility testing of an education program promoting effective parenting habit (Experimental): Parents will receive a series of 6 short videos via Whatsapp
  Interventions: Behavioral: HabitE (effective parenting habit) program (in Brazilian Portuguese)

INTERVENTIONS:
Behavioral: HabitE (effective parenting habit) program (in Brazilian Portuguese) — Parents who enroll in the program will receive a series of 6 videos (~ 7 minutes each), 1 video at a time, generally every 3 days. They will also receive daily written texts, which include implementation tips and an assessment of a target (transition) behavior.

SUMMARY:
This study evaluates the feasibility and preliminary impacts of a new parenting program consisting of a series of educational videos, automatically delivered via a popular texting platform. The program content for the feasibility study is focused on teaching parents strategies to better manage one of the commonly reported challenges that children face, a transition to a non-preferred activity. Parents with young children experiencing behavior difficulties with daily transition routines are invited to participate in the study.

DETAILED DESCRIPTION:
This feasibility study employs a pre-post, open trial design with the primary aim to investigate the feasibility of the automated delivery of parenting educational materials via a widely used texting platform. The training videos demonstrate the applications of antecedent- and reinforcement-based behavior management techniques in a specific situation and encourage parents to build positive parenting habits. The program usability and satisfaction will be assessed through daily interactions of the participants with the program and post-program questionnaires. The study targets parents of children demonstrating behavioral difficulties managing everyday routines at home, while having difficulty accessing traditional forms of psychosocial treatment. In particular, children of ADHD often experience these difficulties, potential participants are informed that the program is for children demonstrating behaviors consistent with ADHD, and ADHD symptoms will be evaluated pre- and post-program participation, although the presence of the disorder will not be required for the program participation. The investigators expect parents to engage well in the program delivered via digital media. Based on the existing literature on the effectiveness of behavior parent training delivered in traditional in-person format, the investigators expect a moderate effect size in the pre-post measures of parenting practices and the child target behavior for this study.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged from 4 to 10 years old
* Parents experiencing behavior difficulties with daily transition routines (parent-report).

Exclusion Criteria:

* Parents that do not have the children living with them at least 5 days per week every week;

  * While participating parents are informed that the program was developed for children demonstrating symptoms of ADHD, the low symptom number will not be used as an exclusion criteria.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of videos viewed | 1 month
  The number of videos viewed (minimum 0, maximum 5) to evaluate participant engagement
Percentage of completed daily ratings | 1 month
  The percentage of completed daily ratings (minimum 0, maximum 17). Parents are asked to provide daily ratings on the degree of success in implementing parenting strategies taught.
Participant satisfaction | 1 month
  The parent-rated satisfaction regarding information presented in the videos. A rating completed after each video viewing using a 4-point scale. Averaged across the ratings completed for the videos viewed. (Minimum 0, maximum 4). Higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Parent-rated child's difficulties with daily transitions | 1 month
  The parent-rated child's difficulties with 9 common daily transitions. Ratings completed before and after the intervention using a 3-point scale. Averaged across the ratings completed for the 9 transitions. Higher scores indicate greater difficulties.
Parent-rated child's impairment related to transition difficulties | 1 month
  The parent-rated level of impairment caused by transition difficulties (1 item). Ratings completed before and after the intervention using a 7 point scale. Higher scores indicate greater impairment.
Inconsistent parenting | 1 month
  Multidimensional Assessment of Parenting Scale (MAPS) Lax Control subscale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 6 items. Lower scores indicate less frequent incidents of inconsistent parenting.
Use of physical control | 1 month
  MAPS Physical Control. Parent ratings completed before and after the intervention using a 5-point scale. Average across 4 items. Lower scores indicate less frequent use of physical disciplines.
Hostility toward child | 1 month
  MAPS Hostility subscale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 7 items. Lower scores indicate less frequent use of hostile reactions during parent-child interactions.
Parent Stress | 1 month
  Parent stress scale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 18 items. Lower scores indicate lower levels of stress.

OTHER OUTCOMES:
ADHD symptoms | 1 month
  Strengths and Weakness of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior Scale (SWAN) inattention and hyperactivity/impulsivity symptoms total. Parent ratings completed before and after the intervention using a 7-point scale. Averaged across 18 items. Higher scores indicate ADHD symptoms more frequently observed.
ODD symptoms | 1 month
  SWAN oppositional/defiant symptoms total. Parent ratings completed before and after the intervention using a 7-point scale. Averaged across 8 items. Higher scores indicate ODD symptoms more frequently observed.
Irritability | 1 month
  Affective Reactivity Index (ARI). Parent ratings completed before and after the intervention using a 3-point scale. Averaged across 6 items. Higher scores indicate irritability more frequently observed.
Proactive parenting | 1 month
  MAPS Proactive Parenting subscale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 6 items. Lower scores indicate less frequent incidents of inconsistent parenting.
Use of positive reinforcement | 1 month
  MAPS Positive Reinforcement subscale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 4 items. Lower scores indicate less frequent use of physical disciplines.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto D'or de Pesquisa e Ensino (IDOR), Brazil, Brazil

IPD SHARING:
Plan to Share IPD: No